CLINICAL TRIAL: NCT05478343
Title: Clinical Trial to Evaluate the Safety and Efficacy of IM21 CAR-T Cells in Patients With Relapsed and Refractory (R/R) Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMCART201909
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM21 CAR-T cells (Experimental)
  Interventions: Biological: IM21 CAR-T cells

INTERVENTIONS:
Biological: IM21 CAR-T cells — IM21 CAR-T cells administrated in a dosage to be selected by physician from a specific range.

SUMMARY:
This is a open-label to determine the efficacy and safety of IM21 CAR-T cells in adult with R/R multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MM with relapsed or refractory disease and have had at least 3 different prior lines of therapy including proteasome inhibitor .
* Evidence of cell membrane BCMA expression.
* Subjects must have measurable disease,including 1) Serum M-protein greater or equal to10 g/L. 2) Urine M-protein greater or equal to 200 mg/24 h. 3)Serum free light chain (FLC) assay: involved FLC level greater or equal to 100 mg/L provided serum FLC ratio is abnormal.
* ≥ 18 years of age at the time of signing informed consent.
* Estimated life expectancy >3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Women of childbearing age who had a negative blood pregnancy test before the start of the trial and agreed to take effective contraceptive measures during the trial period until the last follow-up; male subjects with fertility partners agreed to take effective contraceptive measures during the trial period until the last follow-up.
* Adequate organ function.
* Voluntarily sign informed consent form(s).

Exclusion Criteria:

* Subjects with graft versus host disease and need to use immunosuppressive agents.
* Subjects who had received chemotherapy or radiotherapy within 3 days prior to the blood collection period.
* Use of systemic steroids in combination within 5 days prior to the blood collection period (except for recent or current use of inhaled steroids)
* Subjects who had previously used any gene therapy product.
* Subjects with known central nervous system disease.
* Subjects with plasmacytic leukemia, Wallenian macroglobulinemia, POEMS syndrome, or primary light-chain amyloidosis.
* Subjects had the following cardiac conditions, including but not limited to unstable angina pectoris, myocardial infarction or coronary artery bypass graft in the 6 months prior to enrollment, severe arrhythmias with poor drug control;
* Subjects infected with active HBV or HCV, HIV, syphilis or other untreated active infections;
* Pregnant or lactating women.
* Subjects who have other uncontrolled diseases and are considered by the researchers to be unsuitable to participate in the study.
* Any situation that the researcher believes may increase the risk of subjects or interfere with the results of clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 28 days after CAR-T cell infusion
  Incidence of treatment related AEs
Persistence of CAR-T cells (cell counts and cell percentage in peripheral blood and bone marrow ) | Up to 24 weeks after CAR-T cell infusion
  The persistence over time of CAR T cells in the peripheral blood as determined by flow cytometry and qPCR.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 24 weeks after CAR-T cell infusion
Overall survival (OS) | Up to 24 weeks after CAR-T cell infusion
Minimal residual disease（MRD） | Up to 24 weeks after CAR-T cell infusion
Duration of Response (DOR) | Up to 24 weeks after CAR-T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Yan, M.D., Principal Investigator — First Hospital of China Medical University
Locations (1):
- Hospital of China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Zhou L, Fu W, Wu S, Xu K, Qiu L, Xu Y, Yan X, Zhang Q, Zhang M, Wang L, Hong R, Chang AH, Yu J, Fu S, Kong D, Li L, Wang Y, Li Z, Jiang H, Huang J, Liu Z, Su N, Wei G, Hu Y, Huang H. Derivation and validation of a novel score for early prediction of severe CRS after CAR-T therapy in haematological malignancy patients: A multi-centre study. Br J Haematol. 2023 Aug;202(3):517-524. doi: 10.1111/bjh.18873. Epub 2023 May 16. PMID 37192741